CLINICAL TRIAL: NCT01968954
Title: A Phase 3 Double-blind,Randomized, Placebo-controlled,Parallel-group Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 In Subjects With Primary Hyperlipidemia Or Mixed Dyslipidemia At Risk Of Cardiovascular Events
Brief Title: Randomized Clinical Trial Of Bococizumab (PF-04950615; RN316) In Subjects With Hyperlipidemia Or Mixed Dyslipidemia At Risk Of Cardiovascular Events
Acronym: SPIRE-HR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1481019; 2013-002642-37 (EudraCT Number); SPIRE-HR (Other: Alias Study Number)
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-03

CONDITIONS: Hyperlipidemia
Keywords: mixed dyslipidemia; high risk of cardiovascular events
MeSH Terms: conditions — Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bococizumab (PF-04950615;RN316) (Experimental)
  Interventions: Drug: Bococizumab (PF-04950615;RN316)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bococizumab (PF-04950615;RN316) — 150 mg every 2 weeks, subcutaneous injection, 12 months
  Other Names: RN316
  Arms: Bococizumab (PF-04950615;RN316)
Other: Placebo — subcutaneous injection, every 2 weeks for 12 months
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized study in subjects with high cholesterol receiving highly effective statins to assess the efficacy, safety and tolerability of Bococizumab (PF-04950615;RN316) to lower LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Treated with a statin.
* Fasting LDL-C > 70 mg/dL and triglyceride <=400 mg/dL.
* High or very high risk of incurring a cardiovascular event.

Exclusion Criteria:

* Pregnant or breastfeeding females.
* Cardiovascular or cerebrovascular event of procedures during the past 30 days.
* Congestive heart failure NYHA class IV.
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (103):
- United States (58):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Cardiovascular Associates of the Southeast, LLC, Birmingham, Alabama
  - Southwest Heart Group, Tucson, Arizona
  - ARA-Arizona Research Associates, Tucson, Arizona
  - Diagnamics, Inc., Encinitas, California
  - Encompass Clinical Research North Coast, Encinitas, California
  - MD Studies, Inc., Fountain Valley, California
  - Alliance Research Centers, Laguna Hills, California
  - Prime Care Clinical Research, Laguna Hills, California
  - Providence Clinical Research, North Hollywood, California
  - San Diego Family Care, San Diego, California
  - St. Joseph's Medical Associates, Stockton, California
  - Orange County Research Center, Tustin, California
  - Clinical Research Advantage, Inc./Cassidy Medical Group - Vista, Vista, California
  - Elite Clinical Trials, Wildomar, California
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - Soundview Medical Associates, Norwalk, Connecticut
  - Eastern Research, Inc., Hialeah, Florida
  - East Coast Institute for Research, LLC at Northeast Florida Endocrine & Diabetes Associates, Jacksonville, Florida
  - Care Partners Clinical Research, LLC, Jacksonville, Florida
  - Prestige Clinical Research Center Inc, Miami, Florida
  - Edgewater Medical Research, New Smyrna Beach, Florida
  - Gulfcoast Medical Research Center, LLC, Tampa, Florida
  - Fellows Research Alliance, Inc., Savannah, Georgia
  - SouthCoast Medical Group, Savannah, Georgia
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Comunity Clinical Research Center, Anderson, Indiana
  - American Health Network of Indiana, LLC, Avon, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Internal Medicine Associates, Eunice, Louisiana
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - Allina Health System, dba Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of MN, Lillehei Clinical Trials Unit, Minneapolis, Minnesota
  - Montana Medical Research Inc., Missoula, Montana
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - Radiant Research, Inc, Akron, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - The Office of Daniel G. Williams, MD, Perrysburg, Ohio
  - Great Lakes Medical Research, LLC, Willoughby, Ohio
  - South Oklahoma Heart Research LLC, Oklahoma City, Oklahoma
  - Integrated Medical Research, PC, Ashland, Oregon
  - Columbia Research Group, Inc., Portland, Oregon
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Perelman Center for Advanced Medicine Heart & Vascular Center, Philadelphia, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - Medical Research South,LLC, Charleston, South Carolina
  - Berkeley Family Practice, Moncks Corner, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - 3 rd Coast Research Associates, Corpus Christi, Texas
  - Texas Center For Drug Development, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Utah Cardiology, P.C., Layton, Utah
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
- Australia (3):
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Core Research Group Pty Ltd, Milton, Queensland
  - The Avenue Cardiovascular Centre, St Kilda East, Victoria
- Canada (6):
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Diex Research Montreal Inc., Montreal, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec
  - Medexa Recherche, Victoriaville, Quebec
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Kardiologie a interni lekarstvi, Prague
  - Lekarsky dum Ormiga, Zlín
- Germany (4):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Klinische Forschung Hannover - Mitte GmbH, Hanover
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hong Kong (2):
  - The Chinese University of Hong Kong, Shatin
  - Department of Medicine & Therapeutics-The Chinese University of Hong Kong, Shatin, NT
- Italy (5):
  - IRCCS Ospedale San Raffaele, Milan, MI
  - IRCCS Centro Cardiologico Fondazione Monzino, Milan, MI
  - IRCCS Istituto Auxologico Italiano, Milan, MI
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo, PA
  - Dipartimento di Medicina Interna e Specialita Mediche Policlinico Umberto I, Roma, RM
- Poland (13):
  - SYNEXUS Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Masovian Voivodeship
  - NZOZ Terapia Optima, Katowice, Silesian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Niepubliczny Zaklad Opieki Zdrowotnej CEREO-MED Sp. z o.o., Lodz
  - Medicus w Opolu Sp z o.o., Opole
  - Medicome Sp. z o.o., Oświęcim
  - Synexus Polska Sp. z o.o Oddzial w Poznaniu, Poznan
  - Centrum Medyczne Ogrodowa Sp. z o.o., Skierniewice
  - Centrum Medyczne "SOPMED" Sp. z o.o., Sopot
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - CSK MSW w Warszawie, Klinika Kardiologii Zachowawczej i Nadcisnienia Tetniczego, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
- South Korea (9):
  - The Catholic University of Korea, Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-Do
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Gangnam Sevrance Hospital, Yeonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] McCush F, Wang E, Yunis C, Schwartz P, Baltrukonis D. Anti-drug Antibody Magnitude and Clinical Relevance Using Signal to Noise (S/N): Bococizumab Case Study. AAPS J. 2023 Sep 2;25(5):85. doi: 10.1208/s12248-023-00846-x. PMID 37658997
- [Derived] Chasman DI, Hyde CL, Giulianini F, Danning RD, Wang EQ, Hickling T, Ridker PM, Loomis AK. Genome-wide pharmacogenetics of anti-drug antibody response to bococizumab highlights key residues in HLA DRB1 and DQB1. Sci Rep. 2022 Mar 11;12(1):4266. doi: 10.1038/s41598-022-07997-5. PMID 35277540
- [Derived] Wang EQ, Bukowski JF, Yunis C, Shear CL, Ridker PM, Schwartz PF, Baltrukonis D. Assessing the Potential Risk of Cross-Reactivity Between Anti-Bococizumab Antibodies and Other Anti-PCSK9 Monoclonal Antibodies. BioDrugs. 2019 Oct;33(5):571-579. doi: 10.1007/s40259-019-00375-0. PMID 31529318
- [Derived] Ridker PM, Rose LM, Kastelein JJP, Santos RD, Wei C, Revkin J, Yunis C, Tardif JC, Shear CL; Studies of PCSK9 Inhibition and the Reduction of vascular Events (SPIRE) Investigators. Cardiovascular event reduction with PCSK9 inhibition among 1578 patients with familial hypercholesterolemia: Results from the SPIRE randomized trials of bococizumab. J Clin Lipidol. 2018 Jul-Aug;12(4):958-965. doi: 10.1016/j.jacl.2018.03.088. Epub 2018 Apr 3. PMID 29685591
- [Derived] Ridker PM, Tardif JC, Amarenco P, Duggan W, Glynn RJ, Jukema JW, Kastelein JJP, Kim AM, Koenig W, Nissen S, Revkin J, Rose LM, Santos RD, Schwartz PF, Shear CL, Yunis C; SPIRE Investigators. Lipid-Reduction Variability and Antidrug-Antibody Formation with Bococizumab. N Engl J Med. 2017 Apr 20;376(16):1517-1526. doi: 10.1056/NEJMoa1614062. Epub 2017 Mar 17. PMID 28304227
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481019&StudyName=Randomized%20Clinical%20Trial%20Of%20RN316%20%28PF-04950615%29%20In%20Subjects%20With%20Hyperlipidemia%20Or%20Mixed%20Dyslipidemia%20At%20Risk%20Of%20Cardiovascular%20Events

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received single dose of placebo matched to PF-04950615 subcutaneous injection once in every 2 weeks over a period of 52 weeks. Participants were followed up to 58 weeks.
- PF-04950615 150 mg: Participants received single dose of PF-04950615 150 mg subcutaneous injection once in every 2 weeks over a period of 52 weeks. Participants were followed up to 58 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-04950615 150 mg
Started | 354 | 357
Treated | 353 | 356
Completed | 314 | 314
Not Completed | 40 | 43
Not completed — Adverse Event | 6 | 3
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 20 | 23
Not completed — Other | 7 | 8
Not completed — Protocol Violation | 0 | 1
Not completed — Did not met inclusion criteria | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04950615 150 mg | Total
Number analyzed (Participants) | 354 | 357 | 711
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.7) | 61.1 (10.2) | 61.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 136 | 266
  Male | 224 | 221 | 445

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 329 | 336
percent change | 1.0 (20.89) | -55.6 (29.17)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; LS-mean difference, associated 95% confidence intervals and p values from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region, triglyceride subgroup; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measures (MMRM); Least Square (LS) Mean Difference = -57.0, 95% CI 2-sided [-61.0 to -53.1], Standard Error of Mean 2.00

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified time points for each arm.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 340) | 1.0 (14.85) | -35.1 (19.23)
  Week 24 (n =331, 337) | 3.2 (19.35) | -31.7 (20.47)
  Week 52 (n =313, 315) | 1.8 (18.50) | -27.3 (23.57)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; Week 12: LS-mean difference, associated 95% confidence intervals and p values from an MMRM model with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region, triglyceride subgroup; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -36.2, 95% CI 2-sided [-38.8 to -33.6], Standard Error of Mean 1.33
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; Week 24: LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region, triglyceride subgroup; Test type: Superiority or Other; LS mean difference = -34.7, 95% CI 2-sided [-37.7 to -31.7], Standard Error of Mean 1.52
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; Week 52: LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region, triglyceride subgroup; Test type: Superiority or Other; LS mean difference = -29.0, 95% CI 2-sided [-32.3 to -25.7], Standard Error of Mean 1.69

3. Secondary Outcome: Percent Change From Baseline in Non- High Density Lipoprotein-Cholesterol (Non HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 339) | 1.3 (19.53) | -50.0 (26.28)
  Week 24 (n =329, 336) | 4.7 (27.81) | -46.2 (28.52)
  Week 52 (n =312, 314) | 2.3 (25.22) | -38.9 (33.32)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -51.6, 95% CI 2-sided [-55.2 to -48.1], Standard Error of Mean 1.80
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean Difference = -50.6, 95% CI 2-sided [-54.9 to -46.4], Standard Error of Mean 2.15
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; Week 52:LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region, triglyceride subgroup; Test type: Superiority or Other; LS mean difference = -41.2, 95% CI 2-sided [-45.8 to -36.5], Standard Error of Mean 2.38

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 339) | 0.3 (19.10) | -51.1 (27.62)
  Week 24 (n =331, 335) | 3.5 (22.39) | -47.3 (30.43)
  Week 52 (n =313, 313) | 1.9 (22.25) | -39.1 (33.39)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -51.5, 95% CI 2-sided [-55.1 to -47.9], Standard Error of Mean 1.84
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -50.6, 95% CI 2-sided [-54.6 to -46.6], Standard Error of Mean 2.05
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -40.8, 95% CI 2-sided [-45.2 to -36.3], Standard Error of Mean 2.26

5. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 339) | 4.7 (84.86) | 1.9 (508.44)
  Week 24 (n =331, 336) | 1.9 (51.82) | 4.4 (465.24)
  Week 52 (n =311, 311) | 1.1 (42.47) | 17.3 (562.63)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.860, MMRM; LS mean difference = -2.9, 95% CI 2-sided [-35.4 to 29.5], Standard Error of Mean 16.55
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 2.1, 95% CI 2-sided [-47.2 to 51.4], Standard Error of Mean 25.11
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 12.9, 95% CI 2-sided [-44.5 to 70.4], Standard Error of Mean 29.25

6. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n= 330, 339) | 1.9 (17.24) | 6.6 (14.24)
  Week 24 (n =329, 336) | 1.0 (15.78) | 7.8 (15.91)
  Week 52 (n =312, 314) | 2.0 (15.73) | 5.3 (16.59)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = 4.7, 95% CI 2-sided [2.4 to 7.0], Standard Error of Mean 1.19
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 6.8, 95% CI 2-sided [4.5 to 9.1], Standard Error of Mean 1.18
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 3.3, 95% CI 2-sided [0.9 to 5.8], Standard Error of Mean 1.25

7. Secondary Outcome: Percent Change From Baseline in Fasting Low-Density Lipoprotein-Cholesterol (LDL-C) at Week 12 in Participants With Primary Hyperlipidemia
Description: Participants with primary hyperlipidemia are defined as participants with triglycerides (TG) level less than (<) 200 milligram per decilitre (mg/dL) (2.26 millimoles per litre [mmol/L]) at pre-randomization.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 262 | 266
percent change | 1.5 (20.89) | -56.8 (27.78)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -59.1, 95% CI 2-sided [-63.4 to -54.8], Standard Error of Mean 2.19

8. Secondary Outcome: Percent Change From Baseline in Fasting Low-Density Lipoprotein-Cholesterol (LDL-C) at Week 12 in Participants With Mixed Dyslipidemia
Description: Participants with mixed dyslipidemia are defined as TG level greater than or equal to (>=) 200 mg/dL (2.26 mmol/L) at pre-randomization.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 67 | 70
percent change | -1.0 (20.95) | -50.9 (33.78)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; LS mean difference = -48.7, 95% CI 2-sided [-58.0 to -39.3], Standard Error of Mean 4.72

9. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Week 24 and 52
Time Frame: Baseline, Week 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 24 (n =331, 336) | 6.3 (32.52) | -50.0 (31.36)
  Week 52 (n =311, 313) | 5.2 (29.69) | -40.9 (38.02)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -56.0, 95% CI 2-sided [-60.8 to -51.2], Standard Error of Mean 2.45
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -46.4, 95% CI 2-sided [-51.8 to -41.0], Standard Error of Mean 2.77

10. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 24 and 52 by Triglyceride Cut-off
Description: Percent change from baseline in fasting LDL-C among participants with TG cut-off of <200 mg/dL and >=200 mg/dL (2.26 mmol/L) were reported in this outcome measure.
Time Frame: Baseline, Week 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  TG <200 mg/dL: Week 24 (n =261, 265) | 7.2 (34.38) | -50.8 (30.90)
  TG <200 mg/dL: Week 52(n =243, 248) | 6.2 (29.95) | -41.1 (38.35)
  TG >=200 mg/dL: Week 24(n =70, 71) | 3.0 (24.30) | -46.9 (33.05)
  TG >=200 mg/dL: Week 52(n =68, 65) | 2.0 (28.74) | -40.1 (37.01)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; TG <200 mg/dL (Week 24): LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region; Test type: Superiority or Other; LS mean difference = -57.6, 95% CI 2-sided [-63.1 to -52.0], Standard Error of Mean 2.82
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; TG <200 mg/dL (Week 52): LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region; Test type: Superiority or Other; LS mean difference = -47.7, 95% CI 2-sided [-53.9 to -41.5], Standard Error of Mean 3.16
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; TG >=200 mg/dL (Week 24): LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region; Test type: Superiority or Other; LS mean difference = -49.3, 95% CI 2-sided [-58.9 to -39.8], Standard Error of Mean 4.83
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 150 mg; TG >=200 mg/dL (Week 52): LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region; Test type: Superiority or Other; LS mean difference = -41.2, 95% CI 2-sided [-52.2 to -30.1], Standard Error of Mean 5.60

11. Secondary Outcome: Percent Change From Baseline in Fasting Triglyceride (TG) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 340) | 5.9 (34.90) | -9.4 (42.00)
  Week 24 (n =331, 336) | 7.0 (37.79) | -13.8 (33.24)
  Week 52 (n =313, 315) | 0.6 (38.33) | -9.3 (48.47)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; Week 12: LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region, triglyceride subgroup; Test type: Superiority or Other; LS mean difference = -14.2, 95% CI 2-sided [-19.9 to -8.5], Standard Error of Mean 2.88
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -19.9, 95% CI 2-sided [-25.1 to -14.7], Standard Error of Mean 2.65
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -9.2, 95% CI 2-sided [-15.7 to -2.8], Standard Error of Mean 3.31

12. Secondary Outcome: Percent Change From Baseline in ApolipoproteinA-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 339) | -0.3 (14.05) | 3.7 (12.56)
  Week 24 (n =331, 336) | -0.8 (12.77) | 4.3 (12.25)
  Week 52 (n =313, 313) | 0.4 (13.13) | 3.3 (13.00)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = 3.7, 95% CI 2-sided [1.8 to 5.7], Standard Error of Mean 1.00
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 4.9, 95% CI 2-sided [3.1 to 6.7], Standard Error of Mean 0.91
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 2.6, 95% CI 2-sided [0.7 to 4.6], Standard Error of Mean 0.98

13. Secondary Outcome: Percent Change From Baseline in ApolipoproteinA-II (ApoA-II) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =327, 339) | -1.8 (12.92) | -1.9 (12.10)
  Week 24 (n =331, 335) | -3.7 (14.40) | -1.9 (13.25)
  Week 52 (n =310, 310) | -3.0 (14.76) | -1.6 (12.91)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.1, 95% CI 2-sided [-1.9 to 1.7], Standard Error of Mean 0.93
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = 1.9, 95% CI 2-sided [-0.1 to 3.9], Standard Error of Mean 1.02
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = 1.0, 95% CI 2-sided [-1.0 to 3.1], Standard Error of Mean 1.03

14. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein-Cholesterol (VLDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percent change
  Week 12 (n =330, 340) | 5.9 (34.90) | -9.4 (42.00)
  Week 24 (n =331, 336) | 7.0 (37.79) | -13.8 (33.24)
  Week 52 (n =313, 315) | 0.6 (38.33) | -9.3 (48.47)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS-Mean Difference = -14.2, 95% CI 2-sided [-19.9 to -8.5], Standard Error of Mean 2.88
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -19.9, 95% CI 2-sided [-25.1 to -14.7], Standard Error of Mean 2.65
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -9.2, 95% CI 2-sided [-15.7 to -2.8], Standard Error of Mean 3.31

15. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein-C (LDL-C) at Week 12 by Trigylceride Cut-Off
Description: Absolute change from baseline among participants with TG cut-off of <200 mg/dL and >=200 mg/dL (2.26 mmol/L) were reported in this outcome measure.
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized.'Number of participants analyzed' signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time points for each arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 353 | 357
mg/dL
  TG <200 mg/dL: Baseline (n =282, 282) | 111.2 (31.28) | 112.8 (36.42)
  TG <200 mg/dL: Change at Week12 (n =262, 266) | 0.4 (22.60) | -63.4 (37.38)
  TG >=200 mg/dL: Baseline (n =71, 75) | 126.5 (42.07) | 125.7 (42.10)
  TG >=200 mg/dL: Change at Week 12 (n =67, 70) | -2.6 (26.98) | -63.1 (44.91)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; TG <200 mg/dL (Week 12): LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region; Test type: Superiority or Other; LS mean difference = -64.2, 95% CI 2-sided [-69.1 to -59.2], Standard Error of Mean 2.51
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; TG >=200 mg/dL (Week 12): LS-mean difference, associated 95% confidence intervals with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographical region; Test type: Superiority or Other; LS mean difference = -59.6, 95% CI 2-sided [-71.4 to -47.7], Standard Error of Mean 5.99

16. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =353, 357) | 114.3 (34.22) | 115.5 (37.99)
  Change at Week 12 (n =329, 336) | -0.2 (23.55) | -63.3 (39.00)
  Change at Week 24 (n =331, 336) | 5.5 (33.14) | -56.0 (39.34)
  Change at Week 52 (n =311, 313) | 3.9 (32.17) | -45.9 (46.43)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -63.4, 95% CI 2-sided [-68.0 to -58.8], Standard Error of Mean 2.35

17. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol (TC) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =354, 357) | 186.0 (40.04) | 189.0 (44.68)
  Change at Week 12 (n =330, 340) | 0.6 (27.64) | -66.8 (42.38)
  Change at Week 24 (n =331, 337) | 5.1 (35.83) | -60.1 (43.33)
  Change at Week 52 (n =313, 315) | 1.8 (35.18) | -51.9 (49.68)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -67.1, 95% CI 2-sided [-72.2 to -62.1], Standard Error of Mean 2.59

18. Secondary Outcome: Absolute Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =354, 357) | 137.2 (37.38) | 140.1 (43.48)
  Change at Week 12 (n =330, 339) | 0.3 (26.53) | -69.8 (43.53)
  Change at Week 24 (n =329, 336) | 5.2 (35.91) | -63.6 (44.37)
  Change at Week 52 (n =312, 314) | 1.3 (33.93) | -53.9 (51.10)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -69.7, 95% CI 2-sided [-74.7 to -64.6], Standard Error of Mean 2.57

19. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B (ApoB) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =354, 357) | 94.0 (21.51) | 95.1 (25.57)
  Change at Week 12 (n =330, 339) | -0.5 (17.32) | -47.9 (28.40)
  Change at Week 24 (n =331, 335) | 2.5 (19.87) | -43.9 (29.95)
  Change at Week 52 (n =313, 313) | 0.9 (20.59) | -36.4 (32.23)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -47.3, 95% CI 2-sided [-50.7 to -43.8], Standard Error of Mean 1.74

20. Secondary Outcome: Absolute Change From Baseline in Lipoprotein(a) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =353, 356) | 44.0 (45.93) | 45.1 (52.30)
  Change at Week 12 (n =330, 339) | -0.6 (10.42) | -11.4 (22.19)
  Change at Week 24 (n =331, 336) | -1.2 (12.62) | -10.6 (20.16)
  Change at Week 52 (n =311, 311) | -1.0 (10.71) | -8.6 (23.78)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -10.6, 95% CI 2-sided [-12.9 to -8.3], Standard Error of Mean 1.17

21. Secondary Outcome: Absolute Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =354, 357) | 48.7 (12.52) | 49.0 (13.23)
  Change at Week 12 (n =330, 339) | 0.4 (7.50) | 2.9 (6.92)
  Change at Week 24 (n =329, 336) | -0.0 (7.90) | 3.3 (7.41)
  Change at Week 52 (n =312, 314) | 0.6 (7.59) | 2.1 (8.32)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = 2.4, 95% CI 2-sided [1.4 to 3.5], Standard Error of Mean 0.55

22. Secondary Outcome: Absolute Change From Baseline in Ratio of Fasting Total Cholesterol to High Density Lipoprotein-Cholesterol (TC/HDL-C Ratio) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
ratio
  Baseline (n =354, 357) | 4.0 (1.10) | 4.1 (1.26)
  Change at Week 12 (n =330, 339) | -0.0 (0.71) | -1.6 (1.17)
  Change at Week 24 (n =329, 336) | 0.1 (0.93) | -1.5 (1.21)
  Change at Week 52 (n =312, 314) | 0.0 (0.85) | -1.2 (1.35)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -1.6, 95% CI 2-sided [-1.7 to -1.4], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -1.5, 95% CI 2-sided [-1.7 to -1.4], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -1.2, 95% CI 2-sided [-1.4 to -1.0], Standard Error of Mean 0.08

23. Secondary Outcome: Absolute Change From Baseline in Ratio of Apolipoprotein B to ApolipoproteinA-I (ApoB/ApoA-I Ratio) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
ratio
  Baseline (n =354, 357) | 0.7 (0.18) | 0.7 (0.21)
  Change at Week 12 (n =330, 339) | 0.0 (0.12) | -0.3 (0.21)
  Change at Week 24 (n =331, 335) | 0.0 (0.16) | -0.3 (0.24)
  Change at Week 52 (n =313, 313) | 0.0 (0.14) | -0.3 (0.25)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; LS mean difference = -0.3, 95% CI 2-sided [-0.4 to -0.3], Standard Error of Mean 0.01
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; LS mean difference = -0.3, 95% CI 2-sided [-0.4 to -0.3], Standard Error of Mean 0.01
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; LS mean difference = -0.3, 95% CI 2-sided [-0.3 to -0.2], Standard Error of Mean 0.02

24. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein-Cholesterol (LDL-C) Less Than or Equal to (<=) 100 Milligram Per Deciliter (2.59 Millimoles Per Litre) at Week 12, 24 and 52
Time Frame: Week 12, 24 and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percentage of participants
  Week 12 (n =330, 336) | 41.5 | 87.5
  Week 24 (n =332, 336) | 37.3 | 82.1
  Week 52 (n =312, 313) | 36.9 | 77.3
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; Week 12; Test type: Superiority or Other; Odds Ratio (OR) = 24.0, 95% CI 2-sided [13.86 to 41.64]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; Week 24; Test type: Superiority or Other; Odds Ratio (OR) = 14.8, 95% CI 2-sided [9.32 to 23.56]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; Week 52; Test type: Superiority or Other; Odds Ratio (OR) = 9.8, 95% CI 2-sided [6.36 to 15.24]

25. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein-Cholesterol (LDL-C) Less Than or Equal to (<=) 70 Milligram Per Deciliter (1.81 Millimoles Per Litre) at Week 12, 24 and 52
Time Frame: Week 12, 24 and 52
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
percentage of participants
  Week 12 (n =330, 336) | 5.5 | 76.8
  Week 24 (n =332, 336) | 3.3 | 69.6
  Week 52 (n =312, 313) | 6.4 | 61.7
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 mg; Week 12; Test type: Superiority or Other; Odds Ratio (OR) = 95.2, 95% CI 2-sided [52.09 to 173.91]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 mg; Week 24; Test type: Superiority or Other; Odds Ratio (OR) = 112.2, 95% CI 2-sided [55.81 to 225.52]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 150 mg; Week 52; Test type: Superiority or Other; Odds Ratio (OR) = 29.1, 95% CI 2-sided [17.13 to 49.49]

26. Secondary Outcome: Plasma PF-04950615 Concentrations at Week 12, 24 and 52
Time Frame: Week 12, 24, 52
Population: Analysis set included participants who received at least 1 dose of PF-04950615. Here, 'n' signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | PF-04950615 150 mg
Number analyzed (Participants) | 356
microgram per milliliter
  Week 12 (n =332) | 5.53 (5.666)
  Week 24 (n =327) | 5.36 (6.029)
  Week 52 (n =306) | 4.07 (4.947)

27. Secondary Outcome: Number of Participants With Adverse Events (AEs) Related to Type 1 or 3 Hypersensitivity Reactions and Injection Site Reactions
Description: Type 1 hypersensitivity or allergic reactions were possible in response to any injected protein and included shortness of breath, urticaria, anaphylaxis and angioedema. Type 3 hypersensitivity reactions were similar to Type 1 hypersensitivity reactions but were likely to be delayed from the time of injection and included symptoms such as rash, urticaria, polyarthritis, myalgia's, polysynovitis, fever and if severe then included glomerulonephritis as well. Injection site reactions included injection site bruising, discolouration, erythema, haematoma, haemorrhage, nodule, induration, pain, pruritus and rash. Participants with type 1 or type 3 hypersensitivity reactions and participants with injection site reactions were reported in this outcome measure.
Time Frame: Baseline up to the end of study (up to 58 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 353 | 356
participants
  Type 1 or 3 hypersensitivity reactions | 2 | 1
  Injection site reactions | 5 | 42

28. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (nAb)
Description: Percentage of participants with at least 1 positive ADA titer or 1 positive nAb titer were reported. Participants with their ADA titer >=6.23 were considered to be ADA positive and participants with their nAb titer >=1.58 were considered to be nAb positive.
Time Frame: Baseline up to the end of study (up to 58 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Participants who received at least 1 dose of PF-04950615 were evaluable for this outcome measure. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04950615 150 mg
Number analyzed (Participants) | 352
percentage of participants
  ADA | 44
  nAb | 27

29. Other Pre Specified Outcome: Absolute Change From Baseline in Triglyceride (TG) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =354, 357) | 149.5 (66.83) | 156.2 (78.75)
  Change at Week 12 (n =330, 340) | 3.8 (57.04) | -23.0 (71.52)
  Change at Week 24 (n =331, 336) | 5.0 (64.34) | -28.9 (68.41)
  Change at Week 52 (n =313, 315) | -7.7 (64.14) | -24.3 (82.21)

30. Other Pre Specified Outcome: Absolute Change From Baseline in ApolipoproteinA-I (ApoA-I) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =354, 357) | 147.5 (24.25) | 147.2 (24.96)
  Change at Week 12 (n =330, 339) | -1.2 (19.46) | 4.6 (18.32)
  Change at Week 24 (n =331, 336) | -2.3 (19.33) | 5.6 (17.53)
  Change at Week 52 (n =313, 313) | -0.2 (19.56) | 3.8 (18.86)

31. Other Pre Specified Outcome: Absolute Change From Baseline in ApolipoproteinA-II (ApoA-II) at Week 12, 24 and 52
Time Frame: Baseline, Week 12, 24, 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 mg
Number analyzed (Participants) | 354 | 357
mg/dL
  Baseline (n =353, 356) | 38.1 (6.46) | 38.2 (6.58)
  Change at Week 12 (n =327, 339) | -0.9 (4.95) | -0.9 (4.63)
  Change at Week 24 (n =331, 335) | -1.7 (5.65) | -1.0 (5.07)
  Change at Week 52 (n =310, 310) | -1.5 (5.54) | -0.9 (5.15)

ADVERSE EVENTS:
Time Frame: Baseline up to the end of study (up to 58 weeks)
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonseriousevent during the study.
Arm/Group | Placebo | PF-04950615 150 mg
Serious Adverse Events (participants affected / at risk) | 40/353 | 45/356
Other Adverse Events (participants affected / at risk) | 185/353 | 205/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=353) | PF-04950615 150 mg (N=356)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 2 | 2
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 5
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Retinal aneurysm (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 4
Non-cardiac chest pain (General disorders) | 3 | 2
Pyrexia (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma of sites other than skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/224 | 0/221 — This is gender specific event. The number of participants evaluable for this event are 224 and 221.
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Nerve root compression (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=353) | PF-04950615 150 mg (N=356)
Angina pectoris (Cardiac disorders) | 4 | 5
Palpitations (Cardiac disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 4 | 8
Diarrhoea (Gastrointestinal disorders) | 6 | 12
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 7 | 7
Vomiting (Gastrointestinal disorders) | 5 | 4
Chest pain (General disorders) | 4 | 2
Fatigue (General disorders) | 5 | 7
Injection site bruising (General disorders) | 2 | 5
Injection site erythema (General disorders) | 3 | 9
Injection site haemorrhage (General disorders) | 2 | 4
Injection site pain (General disorders) | 4 | 6
Injection site pruritus (General disorders) | 0 | 4
Injection site reaction (General disorders) | 5 | 42
Non-cardiac chest pain (General disorders) | 5 | 1
Pain (General disorders) | 5 | 0
Acute sinusitis (Infections and infestations) | 3 | 5
Bronchitis (Infections and infestations) | 14 | 13
Cellulitis (Infections and infestations) | 4 | 2
Gastroenteritis (Infections and infestations) | 8 | 2
Herpes zoster (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 7 | 10
Nasopharyngitis (Infections and infestations) | 27 | 26
Pharyngitis (Infections and infestations) | 3 | 6
Pneumonia (Infections and infestations) | 1 | 8
Rhinitis (Infections and infestations) | 1 | 4
Sinusitis (Infections and infestations) | 5 | 10
Upper respiratory tract infection (Infections and infestations) | 19 | 14
Urinary tract infection (Infections and infestations) | 6 | 11
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Fall (Injury, poisoning and procedural complications) | 13 | 10
Muscle strain (Injury, poisoning and procedural complications) | 1 | 5
Alanine aminotransferase increased (Investigations) | 4 | 0
Blood cortisol decreased (Investigations) | 5 | 6
Blood creatine phosphokinase increased (Investigations) | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 6 | 1
Vitamin D decreased (Investigations) | 3 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 5
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 36 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 5
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Dizziness (Nervous system disorders) | 12 | 1
Headache (Nervous system disorders) | 14 | 8
Hypoaesthesia (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 5 | 1
Depression (Psychiatric disorders) | 3 | 6
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3/224 | 1/221 — This is gender specific event. The number of participants evaluable for this event are 224 and 221.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Hypertension (Vascular disorders) | 11 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.